CLINICAL TRIAL: NCT06824155
Title: Phase 0/1 Study of the Safety and Tolerability of 177Lu-RAD202, a Lutetium-177 Radiolabeled Single Domain Antibody Against Human Epidermal Growth Factor Receptor 2 in Patients With Advanced Solid Tumours
Brief Title: HEAT Trial (HER2 Antibody Therapy With Lutetium-177)
Acronym: RAD202
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Radiopharm Theranostics, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAD202.2022.0002
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: HER2 Gene Mutation; Advanced Solid Tumors
Keywords: HER2 positive; Neoplastic disorder; Advanced solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 177Lu-RAD202 (Experimental): Single-arm, open-label study of 177Lu-RAD202 consisting of a Phase 0 Imaging Period (Im) and a Phase 1 Treatment Period (Tr)
  Interventions: Drug: 177Lu-RAD202

INTERVENTIONS:
Drug: 177Lu-RAD202 — 177Lu-RAD202 administered at Imaging (im) and Treatment (tr) doses

SUMMARY:
This is a first-in-human, Phase 0/1, open-label study of177Lu-RAD202 consisting of an Imaging Period with 177Lu-RAD202im(imaging dose) and a Treatment Period with 177Lu-RAD202tr(treatment dose) to determine the recommended dose(s) for future exploration of 177Lu-RAD202 in participants with HER2 expressing advanced solid tumours.

DETAILED DESCRIPTION:
This is a first-in-human, Phase 0/1, open-label study of 177Lu-RAD202 consisting of an Imaging Period with 177Lu-RAD202im (imaging dose) and a Treatment Period with 177Lu-RAD202tr (treatment dose) to determine the recommended dose(s) for future exploration of 177Lu-RAD202 in participants with HER2 expressing advanced solid tumours.

Screening Period: Screening period of up to 4 weeks Phase 0 (Imaging Period): Low dose (10mCi) 177Lu-RAD202 administered on Imaging Day 1 with a follow-up period of up to 2 weeks to assess imaging, safety and dosimetry. Following assessment of the imaging, safety and dosimetry results of the first 3 to 6 participants dosed with 10mCi 177Lu-RAD202im the dose may be increased in subsequent participants, if needed, to improve image quality.

Phase I (Treatment Period): 177Lu-RAD202tr dose escalation

* Treatment Period with each cycle lasting 6 weeks. Extension of the planned dose intervals are possible following discussion and agreement between the Sponsor and Investigator.
* Participants may be treated with multiple cycles as long as they appear to derive clinical benefit as determined by the Investigator and provided adequate clinical safety and organ dosimetry data.
* DLT observation period for 177Lu-RAD202tr is 6 weeks following first injection of 177Lu-RAD202tr.
* Should an alternative treatment schedule be explored, the DLT observation period for 177Lu-RAD202tr at that dose level will be the proposed cycle duration.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years and older.
2. Written, voluntary, informed consent of the participants must be obtained in compliance with institutional, regional, and federal guidelines.
3. Participants with histologically or cytologically confirmed, HER2 positive or HER2-low, advanced solid tumours that are relapsed/refractory, locally advanced not amenable to curative-intent therapy, or metastatic, with documented disease progression during or after their most recent line of anti-cancer therapy. Participants must be refractory to or intolerant of standard of care therapy or have no standard of care therapy available that is likely to provide clinical benefit.

   Participant HER2 positivity is determined by local testing and is defined as a score of 3+ on immunohistochemical analysis IHC), or, defined as a score of 2+ on IHC and positive results on in situ hybridisation (ISH). HER2-low is defined as a score of 1+ on IHC analysis or a score of 2+ on IHC analysis with ISH negative. If the participant tumor's HER2 status is unknown, it may be determined in a pre-screening step whereby the participant is asked to provide written informed consent to have their tumor tissue undergo IHC testing as determined by a validated test (tumor tissue may be obtained from archived samples or from a freshly obtained biopsy).
4. Must have at least 1 measurable target lesion according to RECIST version 1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
6. Participants must have a life expectancy of ≥4 months in the opinion of the Investigator.
7. Women of childbearing potential (WOCBP) must have a negative serum beta-human chorionic gonadotropin (β-hCG) test and must not be breastfeeding. WOCBP are defined as those who are not surgically sterile or post-menopausal. Female participants will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.
8. WOCBP must agree to use a highly effective method of contraception during the study and for 90 days after the last dose of 177Lu-RAD202. Acceptable methods of contraception are described in Section 12.3.3 of the Protocol.
9. Male participants who are able to father a child must agree to avoid impregnating a partner and to adhere to a highly effective method of contraception during the study and for 90 days after the last dose of 177Lu-RAD202. All male participants must agree to not donate sperm during the study and at least 14 days after the last injection of 177Lu-RAD202im and/or 90 days after the last dose of 177Lu-RAD202tr, whichever occurs later. Acceptable methods of contraception are described in Section 12.3.3 of the Protocol.
10. Participants with previously treated brain metastases are eligible to participate if:

    1. They are neurologically and radiologically stable (no evidence of progression by imaging; same imaging modality [magnetic resonance imaging (MRI) or computed tomography (CT) scan] must be used for each assessment),
    2. Do not require steroids to treat associated neurological symptoms, and
    3. Participants have no history of leptomeningeal disease or spinal cord compression.
    4. Participants with active brain metastases untreated with brain-directed therapy such as radiotherapy, are not eligible.
11. For Phase 1 (Treatment Period): Participants must have positive lesion(s) by 177Lu-RAD202im SPECT/CT per central review.

Exclusion Criteria:

1. Participants who have any other known, active malignancy, except for treated cervical intraepithelial neoplasia, or nonmelanoma skin cancer. Participants with a history of malignancies of low recurrence potential who have received curative-intent therapy may be approved on a case-by-case basis in discussion with the study Sponsor, if it is determined not to put the participant at an increased risk of adverse drug effects and/or interfere with the integrity of study outcome.
2. Participants who have any medical condition that would, in the Investigator's judgment, prevent the participant's full participation in the clinical study due to safety concerns or compliance with clinical study procedures such as participants with severe claustrophobia who are unresponsive to oral anxiolytics, participants with low back pain who cannot lie comfortably on an imaging table, participants who are hyperactive or hyperkinetic such that they cannot tolerate lying still for multiple time-point imaging procedures, etc.
3. Residual toxicity Grade ≥ 2 from previously administered therapy (except for alopecia).
4. Inadequate organ functions as reflected in laboratory parameters:

   * Creatinine clearance or Body Surface Area (BSA) adjusted Estimated glomerular filtration rate (eGFR) (calculated using any clinically validated formula, preferably Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI), or measured) < 60 mL/min
   * Platelet count of < 80 x 109/L
   * Absolute neutrophil count (ANC) < 1.5 x 109/L
   * Haemoglobin < 9 g/dL
   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 x upper limit of normal (ULN), or > 5 x ULN for patients with known liver metastases
   * Total bilirubin > 1.5 x ULN, except for participants with documented Gilbert's syndrome who are eligible if total bilirubin ≤ 3 x ULN
   * For participants not taking warfarin or other anticoagulants: international normalized ratio (INR) ≥ 1.5 or prothrombin time (PT) ≥ 1.5 × ULN; and either partial thromboplastin time or activated partial thromboplastin time (PTT or aPTT) ≥1.5 × ULN. Participants taking warfarin must be on a stable dose that results in a stable INR < 3.5. Among participants receiving other anticoagulant therapy, PT or aPTT must be within the intended therapeutic range of the anticoagulant.
5. Significant cardiovascular disease including:

   * Unstable angina and/or myocardial infarction within 6 months prior to screening
   * New York Heart Association Class II or greater congestive heart failure
   * Clinically significant abnormalities in rhythm, conduction, or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block)
   * QT interval corrected for heart rate using Fridericia's formula (QTcF) > 470 msec for females and QTcF > 450 msec for males on screening electrocardiogram (ECG) or congenital long QT syndrome
   * Uncontrolled hypertension
   * Known LVEF < 50%. (LVEF may be performed either by echocardiogram or other appropriate imaging modalities such as nuclear cardiac imaging (MUGA) or MRI).
6. History of uncontrolled allergic reactions and/or have hypersensitivity to anti-HER2 monoclonal antibodies, kanamycin A or aminoglycoside therapies, or other excipients that may induce hypersensitivity
7. Pregnant or lactating women
8. Participants who are receiving any other investigational agents

   The following exclusion criteria applies to participants in Phase 1 (Treatment Period):
9. Received anti-cancer therapy, including chemotherapy, immunotherapy, radiation therapy, biologic, herbal therapy, or any investigational therapy or investigational device, within 28 days (or 5 half-lives for biologic/non-cytotoxic agents, whichever is shorter), prior to the first dose of 177Lu-RAD202tr.
10. Has had or is scheduled to have major surgery ≤ 28 days prior to the first dose of 177Lu-RAD202tr. Surgical procedures not considered to put participants at higher risk of AEs and/or interfere with the integrity of study outcome may be allowed on a case-by-case basis in discussion with the Sponsor.
11. Positive status for human immunodeficiency virus (HIV).
12. Active or chronic hepatitis B or C. Chronic hepatitis B or hepatitis C with undetectable viral loads on stable suppression therapy may be allowed on a case-by-case basis in discussion with study Sponsor.
13. Any medical condition which, in the opinion of the Investigator, places the participant at an unacceptably high risk for toxicities.
14. Any uncontrolled intercurrent illness or clinically significant uncontrolled condition(s), including but not limited to active bacterial, fungal, or viral infections requiring systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Time Activity Curves (TACs) | 72 hours
  Percent of the injected activity vs time for selected organs and tumors
Radiation dosimetry of Lu177-RAD202im | 72 hours
  Absorbed radiation doses of 177Lu-RAD202im in critical organs (e.g., kidneys, bone marrow)
Safety and tolerability of a single dose of 177Lu-RAD202tr | 6 weeks
  The properties, incidence, nature and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) per Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Recommended dose(s) of 177Lu-RAD202tr for future exploration | 6 weeks
  Incidence of dose-limiting toxicities (DLTs) during the first 6 weeks following 177Lu-RAD202tr injection cycle of treatment
Pharmacokinetics of 177Lu-RAD202im | 72 hours
  Half-life of 177Lu-RAD202im in blood
Biokinetics of 177Lu-RAD202im | 72 hours
  Time-integrated activity coefficients of 177Lu-RAD202im in organs and tumor lesions

SECONDARY OUTCOMES:
Safety and tolerability of 177Lu-RAD202im | 6 weeks
  The properties, incidence, nature and severity of AEs and SAEs per Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Recommended dose(s) of 177Lu-RAD202im for future exploration | 2 weeks
  Incidence of dose-limiting toxicities (DLTs) in the first 2 weeks following 177Lu-RAD202im injection
Preliminary antitumor activity of 177Lu-RAD202tr | Up to 30 weeks
  Objective response rates (ORR) as assessed by RECIST v1.1
Radiation dosimetry of 177Lu-RAD202tr | 72 hours
  Absorbed radiation doses of 177Lu-RAD202tr in critical organs (e.g., kidneys, bone marrow)

OTHER OUTCOMES:
Level of agreement between 177Lu-RAD202im and standard of care imaging | Up to 30 weeks
  Standard of care imaging may include but is not limited to 18F-FDG-PET, CT-scan and/or 99mTc-MDP-bone
Effect of 177Lu-RAD202im and 177Lu-RAD202tr on tumor markers | Up to 30 weeks
  Circulating tumor DNA

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Nepean Hospital, Kingswood, New South Wales
  - Macquarie University Hospital, Macquarie Park, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - St Vincents Hospital, Melbourne, Fitzroy, Victoria
  - GenesisCare Murdoch, Murdoch, Western Australia

IPD SHARING:
Plan to Share IPD: No